CLINICAL TRIAL: NCT01134848
Title: A Randomised, Double Blind Cross-over Study of Serial MRCP Following Morphine-neostigmine and Secretin Provocation in Healthy Volunteers
Brief Title: A Study of Serial Magnetic Resonance Cholangiopancreatography (MRCP) Following Morphine-neostigmine and Secretin Provocation in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Paul Cartledge, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: C/10/2007
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Sphincter of Oddi Dysfunction
Keywords: Bile ducts; Sphincter of Oddi; Pancreatic ducts
MeSH Terms: conditions — Sphincter of Oddi Dysfunction | interventions — Morphine; Neostigmine; Saline Solution; Secretin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine-neostigmine (Active Comparator)
  Interventions: Drug: Morphine; Drug: Neostigmine; Drug: 0.9% saline
- Secretin (Active Comparator)
  Interventions: Drug: Secretin; Drug: 0.9% saline

INTERVENTIONS:
Drug: Morphine — 10mg IM
  Arms: Morphine-neostigmine
Drug: Neostigmine — 1mg IM
  Arms: Morphine-neostigmine
Drug: 0.9% saline — 0.1 ml/kg
  Arms: Morphine-neostigmine
Drug: Secretin — 1 unit/kg IV
  Arms: Secretin
Drug: 0.9% saline — 1ml IM
  Arms: Secretin

SUMMARY:
The sphincter of Oddi is a circular band of muscle which controls the flow of pancreatic juices and bile into the small intestine. Abnormal function of the Sphincter of Oddi, known as Sphincter of Oddi dysfunction (SOD), can lead to recurrent episodes of abdominal pain. Making a diagnosis of SOD is difficult and is currently achieved using an invasive pressure test. This pressure test is associated with some adverse effects including inflammation of the pancreas gland. We are investigating an alternative test in which medication is given to provoke spasm of the sphincter. Following provocation, blood can be sampled to detect changes in blood composition and changes in sphincter anatomy can be evaluated using specialized imaging techniques.

Our aim is to study and compare the effects of two provocation medications (morphine-prostigmine and secretin) on biliary and pancreatic ductal anatomy, using dynamic serial MRCP in healthy volunteers.

Our hypothesis is that morphine-neostigmine provocation results in greater changes in biliary and pancreatic ductal anatomy when assessed using dynamic serial MRCP.

DETAILED DESCRIPTION:
The sphincter of Oddi (SO), which encases the distal common bile duct (CBD) and pancreatic duct (PD), comprises a fibromuscular complex to control the flow of biliary and pancreatic secretions into the duodenum. Aberrant function of the SO, known as Sphincter of Oddi dysfunction (SOD), can lead to recurrent episodes of biliary or pancreatic type pain. Both surgical sphincteroplasty and endoscopic sphincterotomy can improve symptoms in some patients who are suspected to have SOD. However, poor results are obtained in a significant proportion reflecting the difficulties in achieving an accurate diagnosis and also in selecting those patients likely to benefit from these procedures. A number of investigative modalities have been employed in the assessment of SOD. Of the available diagnostic tests sphincter of Oddi manometry (SOM) is considered the gold standard, but is associated with a high rate of post procedure morbidity including pancreatitis and biliary sepsis.

It is therefore unsurprising that attention has focussed on non-invasive diagnostic tests. Developments in magnetic resonance cholangiopancreatography (MRCP) have allowed for the detailed non-invasive assessment of biliary and pancreatic ductal morphology and can be used in conjunction with intravenous secretin provocation (ss-MRCP). Evaluations of this technique have so far been disappointing, demonstrating only a modest concordance with SOM in patients suspected with SOD.

The morphine-prostigmine provocation test (Nardi test) has previously been utilised as a screening test in patients with symptoms suggestive of SOD. It is performed by giving an intramuscular injection of morphine 10mg and prostigmine 1mg, with a positive test indicated by the reproduction of pain or a fourfold increase in either serum amylase or lipase levels. As enzymatic changes have been shown to occur in healthy subjects and in those with irritable bowel syndrome, the test has largely fallen out of favour. However, a recent publication has suggested morphine used as a pharmacological provocation agent can improve ductal distension and aid the differentiation of pancreaticobiliary variants on MRCP. To date this has not been investigated in a randomised or blinded study and we have therefore proposed to examine the effects of morphine-neostigmine and secretin provocation on gallbladder volume and biliary and pancreatic ductal morphology in healthy volunteers using serial MRCP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy age matched and sex matched volunteers
* No history of chronic abdominal pain
* No previous abdominal surgery
* No history suggestive of gastrointestinal motility disorders
* No history of regular medication or substance abuse

Exclusion Criteria:

* Acute illness within preceding 6 weeks
* Participation in another study within 3 months
* Allergy to morphine or neostigmine
* Pregnancy
* Refusal to consent to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Serum amylase (U/L) | 0, 60, 120, 180 and 240 minutes
Serum lipase (U/L) | 0, 60, 120, 180 and 240 minutes
Liver function tests | 0, 60, 120, 180 and 240 minutes

SECONDARY OUTCOMES:
Pancreatic duct diameter (mm) | 0, 5, 30, 60, 90, 120, 150 and 180 minutes
Pancreatic duct length (mm) | 0, 5, 30, 60, 90, 120, 150 and 180 minutes
Common bile duct diameter (mm) | 0, 5, 30, 60, 90, 120, 150 and 180 minutes
Gallbladder volume (mm3) | 0, 5, 30, 60, 90, 120, 150 and 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Lobo, MBBS DM FRCS, Principal Investigator — University of Nottingham; Abeed Chowdhury, MB ChB BSc MRCS, Study Director — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom